CLINICAL TRIAL: NCT04402398
Title: Psychometric Properties of a Mobile Application in Pressure Ulcers for Patients With Spinal Cord Injuries (SCI)
Brief Title: Psychometric Properties of a Mobile Application
Acronym: IMITO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0280
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Spinal Cord Injuries
Keywords: Pressure ulcer; validity of measures
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current methods to assess superficial size and area of pressure ulcers are either time-consuming (using Transparency Tracings techniques), costly (computers, softwares), or necessitating to touch the patient's skin (using commun rulers).

A free smartphone application (for IOS or Android) has recently been developed to measures skin lesions. It is called imitoMeasure. It does not require any contact with the patient. A photograph is taken with the smartphone, the limits of the lesion is then drawn with the health carers' finger on the phone's screen. The application computes the length, width and surface of the ulcer.

This technique has not yet been validated, although it has been used to measure various types of skin lesions.

The objective of this study is to validate this measurement technique on a sample of pressure ulcer in a population of patients with spinal cord injury (SCI). Reliability is assessed by comparison to the currently most frequently used techniques (Transparency Tracings and ruler-based), and fiability is assessed by intra-rater and inter-rater correlations.

imitoMeasure is a new smartphone application to measure wounds size. The present study assesses validity of the measure against common measures (ruler-based and transparency tracings), and the inter- and intra-rater reliability.

ELIGIBILITY:
Inclusion criteria:

* complete or incomplete spinal cord injury, all delays or aetiologies
* presence of one or more pressure ulcers stade II to IV
* adults

Exclusion criteria:

* refusal to participate
* local infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients, providing consent for study, with complete or incomplete spinal cord injury, with pressure ulcers requiring hospital follow-up (lesion stade II to IV), followed at Centre Mutualiste Propara, rehabilitation centre, Montpellier, France
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Correlation of imitoMeasure of ulcers' surface to transparency tracing surface measure | immediately upon first assessment of patients
  Correlation of imitoMeasure of ulcers' surface to transparency tracing surface measure

SECONDARY OUTCOMES:
Correlation of imitoMeasure of ulcers' surface to ruler-based surface measure | immediately upon first assessment of patients
  Correlation of imitoMeasure of ulcers' surface to ruler-based surface measure
inter-rater and intra-rater validity of imitoMeasure | immediately upon first assessment of patients
  inter-rater and intra-rater validity of imitoMeasure
Correlation of imitoMeasure of length and width of ulcers to ruler-based measures | immediately upon first assessment of patients
  Correlation of imitoMeasure of length and width of ulcers to ruler-based measures

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LAFFONT, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Do Khac A, Jourdan C, Fazilleau S, Palayer C, Laffont I, Dupeyron A, Verdun S, Gelis A. mHealth App for Pressure Ulcer Wound Assessment in Patients With Spinal Cord Injury: Clinical Validation Study. JMIR Mhealth Uhealth. 2021 Feb 23;9(2):e26443. doi: 10.2196/26443. PMID 33620327